CLINICAL TRIAL: NCT00489242
Title: PREDICT Trial: Prediction of CK-MB Release During Otherwise Successful Stenting Procedure Correlating With Indicators of Microvascular Obstruction
Brief Title: Prediction of CK-MB Release During Otherwise Successful Stenting Procedure
Acronym: PREDICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H4S-MC-X022; GCO #: 02-1162
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Procedure: Procedure / Percutaneous angioplasty

SUMMARY:
Aims of this study will be to assess the difference in CFV/CFR (Coronary flow velocity/reserve) in diabetic vs. non-diabetic patients and to correlate CK-MB, TnI and HsCRP release after otherwise successful coronary stenting.

DETAILED DESCRIPTION:
Post-procedure CK-MB and troponin I (TnI) and HsCRP elevation, in the absence of obvious procedural events, is most likely caused by distal micro-thromboembolism of platelet aggregates and atheromatous debris causing microvascular bed obstruction. This, in turn, will result in lower coronary flow reserve and regional left ventricular (LV) dysfunction. Therefore, patients with normal CFV/CFR (coronary flow velocity/reserve) by Doppler wire and FFR (fractional flow reserve) by flow wire should have no peri-procedural CK-MB, TnI elevation as compared to patients with peri-procedural CK-MB and TnI elevation where all markers of microcirculation will be reduced. This observation will have a prognostic value at short and long-term. This study may also have clinical implications for patients with intra-coronary stenting and normal microvascular parameters post PCI that these patients may be discharged early while others may need to be monitored in-hospital for an extended period of time.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Stable patients who will undergo PCI (intent to stent)
* Patients with de novo type B2/C lesions of native coronary vessels

Exclusion Criteria:

* Patients with acute myocardial infarction (Q wave or non-Q wave with CK-MB 5 times above the upper normal [80 U/L] within 72 hours)
* Patients who are in cardiogenic shock
* Patients with restenotic lesions
* Patients with type A and type B1 lesions of native coronary vessels
* Patients who require use of atherectomy devices for PCI
* Patients who have elevated CK-MB (>16 U/L) or TnI (>2ng/L) at baseline
* Patients who receive tirofiban or eptifibatide infusion within 24 hours of PCI
* Patients with known allergy to abciximab and adenosine
* Patients with platelet count <100,000 cell/mm3
* Patients who have co-morbidity which reduces life expectancy to one year
* Patients who are currently participating in another investigational drug/device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-08; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
To assess the difference in CFV/CFR (coronary flow velocity/coronary flow reserve) in diabetic versus non-diabetic patients and to correlate CK-MB, TnI and HsCRP release after otherwise successful coronary stenting.

SECONDARY OUTCOMES:
Correlation of CK-MB, Troponin-I and HsCRP release with CFR<2.0, FFR<0.8 in diabetic vs non-diabetic group. Evaluation of 30-day Major Adverse Cardiac Events (MACE) defined as death, MI, or urgent revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Annapoorna S. Kini, MD,, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States